CLINICAL TRIAL: NCT01431937
Title: A Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Repeat Ascending Doses of GSK2018682 (S1P1 Agonist) in Healthy Volunteers
Brief Title: Assessment of Repeat Ascending Doses of GSK2018682 in Healthy Volunteers
Acronym: P1A114347
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 114347
Record Dates: First submitted 2011-08-11; First posted 2011-09-12 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — GSK2018682

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2018682 (Active Comparator): Active Drug
  Interventions: Drug: GSK2018682
- Placebo Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2018682 — Active Drug
  Arms: GSK2018682
Drug: Placebo — Placebo
  Arms: Placebo Control

SUMMARY:
The study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of repeat ascending doses of GSK2018682. The study will also provide further evidence of the potential therapeutic dose-range by measuring the inhibitory effect of GSK2018682 on Absolute Lymphocyte Counts (ALC).

DETAILED DESCRIPTION:
The study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of repeat ascending doses of GSK2018682. The study will also provide further evidence of the potential therapeutic dose-range by measuring the inhibitory effect of GSK2018682 on Absolute Lymphocyte Counts (ALC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Females must be of non-childbearing potential.
* BMI within the range 19 - 29 kg/m2 (inclusive).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Were participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Other exclusion criteria to be detailed at the time of physical screening by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10-10 (Actual); Primary Completion 2011-03-29 (Actual); Study Completion 2011-03-29 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of repeat oral doses of GSK2018682 in healthy volunteers (males and females of non-childbearing potential) | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  Adverse event monitoring, Laboratory parameters (haematology, clinical chemistry, urinalysis), Ophthalmic examination
To investigate effects of repeat oral doses of GSK2018682 on heart rate and blood pressure in healthy volunteers | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  12-lead ECG, Telemetry ECG, Holter ECG, Vital signs (systolic and diastolic blood pressure, heart rate, respiratory rate, body temperature), Ambulatory blood pressure monitoring
To investigate effects of repeat oral doses of GSK2018682 on lung function in healthy volunteers | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  FEV1 obtained via spirometry
To investigate the pharmacokinetics of repeat oral doses of GSK2018682 in healthy volunteers | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  Peak blood concentration, Time of peak blood concentration, Area under the blood concentration-time curve over the 24-hour dose interval and area under the blood concentration-time curve from time-zero extrapolated to infinite time, Accumulation ratio, Terminal half-life, Apparent oral clearance, Through concentration
To characterize the metabolism of GSK2018682 | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  GSK2018682 bile metabolites, GSK2018682 whole blood metabolites
Evaluate the effect of repeat oral doses of GSK2018682 on lymphocytes in healthy volunteers | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  % Change from baseline in absolute lymphocyte counts (ALC), % Change from baseline in subsets CD3+ [CD4+ and CD8+], CD19+, CD16+/CD56+ counts, % Change from baseline in further defined functional T cell subsets (naïve, central memory, effector memory and regulatory T cells)
To explore the PK/PD relationship between blood concentrations and changes in vital signs and ECG parameters | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  PK/PD model with parameters of the models will be determined that best describe the relationship between blood concentrations of GSK2018682 and vital signs and ECG parameters
To explore the PK/PD relationship between blood concentrations of GSK2018682 and reduction in lymphocyte counts | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 13 weeks
  PK/PD model with parameters of the models will be determined that best describe the relationship between blood concentrations of GSK2018682 and reduction ALC and subset counts CD3+ [CD4+ and CD8+], CD19+, CD16+/CD56+ and further defined functional T cell subsets (naïve, central memory, effector memory and regulatory T cells)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Australia (3):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114347 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114347?search=study&search_terms=114347#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register